CLINICAL TRIAL: NCT03557931
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Parallel-group Study to Assess the Safety and Efficacy of ASP4345 as Add-on Treatment for Cognitive Impairment in Subjects With Schizophrenia on Stable Doses of Antipsychotic Medication
Brief Title: A Study to Assess the Safety and Efficacy of ASP4345 as Add-on Treatment for Cognitive Impairment in Subjects With Schizophrenia on Stable Doses of Antipsychotic Medication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4345-CL-0015
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2020-10-27 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
Keywords: aripiprazole; ziprasidone; lurasidone; schizophrenia; ASP4345; quetiapine; olanzapine; brexpiprazole; risperidone; paliperidone
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Quetiapine Fumarate; Olanzapine; ziprasidone; Aripiprazole; brexpiprazole; Paliperidone Palmitate; Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ASP4345 50 milligram (mg) (Experimental): Participants on stable doses of antipsychotic medication received ASP4345 50 mg, capsules, orally, once daily for 12 weeks.
  Interventions: Drug: ASP4345; Drug: risperidone; Drug: quetiapine; Drug: olanzapine; Drug: ziprasidone; Drug: aripiprazole; Drug: brexpiprazole; Drug: paliperidone; Drug: lurasidone
- ASP4345 150 mg (Experimental): Participants on stable doses of antipsychotic medication received ASP4345 150 mg, capsules, orally, once daily for 12 weeks.
  Interventions: Drug: ASP4345; Drug: risperidone; Drug: quetiapine; Drug: olanzapine; Drug: ziprasidone; Drug: aripiprazole; Drug: brexpiprazole; Drug: paliperidone; Drug: lurasidone
- Placebo (Placebo Comparator): Participants on stable doses of antipsychotic medication received ASP4345 placebo matching capsules, orally, once daily for 12 weeks.
  Interventions: Drug: placebo; Drug: risperidone; Drug: quetiapine; Drug: olanzapine; Drug: ziprasidone; Drug: aripiprazole; Drug: brexpiprazole; Drug: paliperidone; Drug: lurasidone

INTERVENTIONS:
Drug: ASP4345 — oral administration
  Arms: ASP4345 150 mg; ASP4345 50 milligram (mg)
Drug: placebo — oral administration
  Arms: Placebo
Drug: risperidone — oral or depot administration
  Other Names: Risperdal
Drug: quetiapine — oral administration
  Other Names: Seroquel
Drug: olanzapine — Oral or depot administration
  Other Names: Zyprexa
Drug: ziprasidone — Oral or depot administration
  Other Names: Geodon
Drug: aripiprazole — Oral or depot administration
  Other Names: Abilify
Drug: brexpiprazole — Oral administration
  Other Names: Rexulti
Drug: paliperidone — Oral or depot administration
  Other Names: Invega
Drug: lurasidone — Oral administration
  Other Names: Latuda

SUMMARY:
The purpose of this study was to evaluate the efficacy of ASP4345 on cognitive impairment compared to placebo using change from baseline in MATRICS Consensus Cognitive Battery (MCCB) neurocognitive composite score (excluding social cognition domain). The primary estimand used a Hypothetical Strategy and compared participants as though the participant had continued on the assigned treatment and to evaluate the safety and tolerability of ASP4345 compared to placebo. This study also evaluated the effects of ASP4345 compared to placebo on functional capacity using the University of California San Diego Performance-based Skills Assessment-2 Extended Range (UPSA-2-ER) total score and evaluated the pharmacokinetic profile of ASP4345.

DETAILED DESCRIPTION:
Participants received oral doses of ASP4345 or matching placebo QD (once daily) for 12 weeks. All participants were administered the first dose of blinded study drug at the site following randomization and provided with web-based applications that provided supplemental cognitive training and recorded treatment compliance. Participants returned to the clinic weekly for safety, efficacy, and/or pharmacokinetic procedures. Participants continued the participant's antipsychotic treatment for the entire study and were followed for 14 days after the participant's last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition criteria and confirmed by the Mini-International Neuropsychiatric Interview version 7.02
* Subject has a stable clinical course as suggested by the following:

  * no psychiatric hospitalization within the last 4 months,
  * no symptom-related changes in psychotropic medications (as defined in the concomitant medication section) within 4 weeks prior to baseline for oral medications and within 2 months for depot medications,
  * and core positive symptoms no worse than moderate in severity and no evidence of a current severe major depressive episode (moderately severe depression is allowed)
* Subject has a stable living situation
* Subject's extrapyramidal symptoms are no worse than mild in severity
* Subject must be in ongoing maintenance (i.e., at least 4 weeks prior to day 1 for oral medications and within 2 months for depot medications) on up to 2 antipsychotic therapies (oral or depot) other than clozapine
* Subject has a body mass index range of 18.5 to 45.0 kg/m2
* Female subject must either:

  * Be of nonchildbearing potential:
  * Postmenopausal (defined as at least 1 year without menses) prior to screening or
  * Documented as surgically sterile
* Or, if of childbearing potential

  * Agrees not to try to become pregnant during the study and for 28 days after the final study drug administration
  * And has a negative blood pregnancy test at screening and a negative urine pregnancy test at day 1,
  * and if heterosexually active, agrees to consistently use 1 form of highly effective birth control starting at screening and throughout the study period and for 28 days after the final study drug administration
* Female subjects must agree not to breastfeed starting at screening and throughout the study period, and for 28 days after the final study drug administration
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration
* A sexually active male subject with female partner(s) who is of childbearing potential is eligible if:

  * Agrees to use male condom starting at screening and throughout the study period, and for 28 days after the final study drug administration
* Male subject must not donate sperm starting at screening and throughout the study period, and for 28 days after the final study drug administration
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or time partner is breastfeeding throughout the study period and for 90 days after the final study drug administration
* Subject agrees not to participate in another interventional study while participating in the present study, defined as signing the informed consent form until completion of the last study visit
* Subject has a negative urine drug screen for drugs of abuse at screening and day 1, excluding cannabis and documented prescribed benzodiazepines

Exclusion Criteria:

* Subject has a known or suspected hypersensitivity to ASP4345 or any components of the formulation
* Subject has had previous exposure with ASP4345
* Subject has a history of suicide attempt or suicidal behavior within 1 year prior to screening or has any suicidal ideation that meets criteria at a level of 4 or 5 by using the Columbia Suicide Severity Rating Scale (C-SSRS) or who is at significant risk to commit suicide
* Subject has any clinically significant liver chemistry test result (aspartate aminotransferase [AST], alanine aminotransferase [ALT], total bilirubin [TBL]) or a result > 1.5 times above the upper limit of normal (ULN) at screening or repeated within

  1 week prior to potential randomization (day 1). In such a case, the assessment may be repeated once
* Subject has any history or evidence of any clinically significant allergic, cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, history of seizure disorder, renal and/or other major disease or malignancy
* Subject has any clinically significant abnormality of the physical examination, electrocardiogram (ECG) and clinical laboratory tests at screening or at admission to the study (day 1)
* Subject has known kidney disease and a glomerular filtration rate (GFR) < 60 mL/min per meter squared at screening and subjects will be discontinued from treatment only for decreases in the GFR that are clinically relevant
* Subject has a resting systolic blood pressure > 180 mmHg or < 90 mmHg, and a resting diastolic blood pressure > 100 mmHg at screening. These assessments may be repeated once, after a reasonable time period, at the investigator's discretion (but within the screening period)
* Subject has a mean corrected QTcF > 450 msec (for male subjects) and > 470 msec (for female subjects) at screening or at randomization. If the mean QTcF exceeds the limits above, one additional triplicate ECG can be taken on day 1
* Subject has a history in the 6 months prior to screening of consuming more than 14 units of alcoholic beverages per week for males and more than 7 units of alcoholic beverages per week for females. (Note 1 unit = 12 ounces of beer, 4 ounces of wine, or 1 ounce of spirits)
* Subject is currently using prohibited medications and is unable to washout, including over-the-counter products and agrees not to consume grapefruit and/or grapefruit juice
* Subject is currently using clozapine for treatment of schizophrenia
* Subject has a positive test for hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (immunoglobulin M) (anti-HAV [IgM]) or hepatitis C virus antibodies (anti- HCV) at Screening or has history of a positive test for human immunodeficiency virus type 1(HIV-1) and/or type 2 (HIV-2)
* Subject who has had electroconvulsive therapy within the 6 months prior to screening.
* Subject has a history of head injury with clinically significant sequelae, including loss of consciousness for 1 hour or greater
* Subject has received investigational study drug within 28 days or 5 half-lives, whichever is longer, prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 233 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director, Study Director — Astellas Pharma Global Development
Locations (27):
- United States (27):
  - CNS Research Science, Inc., Cerritos, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Synergy East, Lemon Grove, California
  - Pacific Research Partners, LLC, Oakland, California
  - California Neuropsychopharmacology Clinical Research Institute-LA, LLC, Pico Rivera, California
  - California Neuropsychopharmacology Clinical Research Institute, LLC (CNRI-San Diego), San Diego, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Sharp Mesa Vista Hospital, San Diego, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Radiant Research, Inc., Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Alam Medical Research Inc., Chicago, Illinois
  - Uptown Research Institute, Chicago, Illinois
  - Michigan Clinical Research Institute PC, Ann Arbor, Michigan
  - Cherry Street Services, Inc., Grand Rapids, Michigan
  - Arch Clinical Trials, LLC, St Louis, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Albuquerque Neuroscience Inc., Albuquerque, New Mexico
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - CNS Research Science, Inc., Jamaica, New York
  - New York State Psychiatric Institute, New York, New York
  - Manhattan Psychiatric Center's 125th Street Clinic, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Desai A, Benner L, Wu R, Gertsik L, Uz T, Marek GJ, Zhu T. Pharmacokinetics of ASP4345 from Single Ascending-Dose and Multiple Ascending-Dose Phase I Studies. Clin Pharmacokinet. 2021 Jan;60(1):79-88. doi: 10.1007/s40262-020-00911-0. PMID 32533536
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=404

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were 18 to 55 years of age (inclusive at screening) with stable schizophrenia or schizoaffective disorder with mild extrapyramidal symptoms on up to 2 antipsychotic therapies and who met inclusion criteria and none of the exclusion criteria were enrolled.
Groups:
- ASP4345 50 Milligrams (mg): Participants on stable doses of antipsychotic medication received ASP4345 50 mg, capsules, orally, once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | ASP4345 50 Milligrams (mg) | ASP4345 150 mg
Started | 100 | 65 | 68
Completed | 69 | 46 | 55
Not Completed | 31 | 19 | 13
Not completed — Adverse Event | 4 | 6 | 1
Not completed — Lost to Follow-up | 4 | 4 | 1
Not completed — Protocol Violation | 1 | 4 | 1
Not completed — Withdrawal by Subject | 14 | 0 | 7
Not completed — Miscellaneous | 8 | 5 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) analysis set consisted of all participants who were randomized into the study.
Groups:
- ASP4345 50 mg: Participants on stable doses of antipsychotic medication received ASP4345 50 mg, capsules, orally, once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | ASP4345 50 mg | ASP4345 150 mg | Total
Number analyzed (Participants) | 100 | 65 | 68 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (9.1) | 42.7 (9.2) | 42.8 (9.9) | 42.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 20 | 70
  Male | 73 | 42 | 48 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 3 | 4 | 21
  Not Hispanic or Latino | 86 | 62 | 64 | 212
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 2 | 1 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 72 | 48 | 47 | 167
  White | 24 | 14 | 17 | 55
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
MATRICS Consensus Cognitive Battery (MCCB) Neurocognitive Composite Score [Mean (Standard Deviation); unit: T-score] — The MCCB is a cognitive battery to assess 7 domains recommended by the MATRICS initiative (ie, working memory, verbal learning, speed of processing, attention/vigilance, visual learning, social cognition, reasoning and problem solving). The MCCB neurocognitive composite score is a standardized mean of the six domain scores (excluding social cognition). Raw scores are converted to age and sex adjusted t-scores which are standardized to normative data, and have a mean of 50 and standard deviation of 10 in the general healthy population. A higher score indicates less impairment. Population: ITT population with available data at baseline.
  T-score
    number analyzed (Participants) | 99 | 65 | 68 | 232
    (all) | 32.6 (13.3) | 34 (10.7) | 33.7 (12.3) | 33.3 (12.3)
UPSA-2-ER Total Score [Mean (Standard Deviation); unit: units on a scale] — The University of California San Diego Performance-based Skills Assessment-2 Extended Range (UPSA-2-ER) assesses the functional abilities of the participant with schizophrenia in 6 domains: household management, communication, financial skills, transportation, comprehension/planning and medication management. The UPSA-2-ER total score has a range from 0 to 105. A higher score indicates less impairment. Population: ITT population with available data at baseline.
  units on a scale
    number analyzed (Participants) | 82 | 59 | 63 | 204
    (all) | 74.4 (16.7) | 80.2 (13.2) | 78.1 (15.5) | 77.2 (15.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12/End of Treatment (EoT) in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Neurocognitive Composite Score
Description: The MCCB is a cognitive battery to assess 7 domains recommended by the MATRICS initiative (i.e., working memory, verbal learning, speed of processing, attention/vigilance, visual learning, social cognition, reasoning and problem solving). The MCCB neurocognitive composite score is a standardized mean of the six domain scores (excluding social cognition). Raw scores are converted to age and sex adjusted t-scores which are standardized to normative data, and have a mean of 50 and standard deviation of 10 in the general healthy population. A higher score indicates less impairment.
Time Frame: Baseline and week 12/end of treatment (EoT)
Population: The full analysis set (FAS) consisted of all participants who were randomized and received at least 1 dose of study drug and had at least 1 postbaseline MCCB measurement. FAS population with available data at baseline and week12/EoT.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | ASP4345 50 mg | ASP4345 150 mg
Number analyzed (Participants) | 67 | 45 | 51
T-score | 1.15 (0.65) | 1.34 (0.79) | 0.87 (0.75)
Statistical Analysis 1: Comparison: Placebo vs ASP4345 50 mg; Mixed model repeated measures (MMRM) analysis model is performed with change from baseline (least square (LS) Mean estimate for observed value from separate model using observed values) at week 12 as response; treatment, site (pooled where necessary), visit, treatment*visit, and visit*baseline as fixed effects, and baseline as a covariate; Test type: Superiority; p = 0.858, MMRM Method; LS Mean Difference = 0.18, 90% CI 2-sided [-1.51 to 1.88], Standard Error of Mean 1.02; Cohen's d Effect Size was defined as: (t-value for the least squares mean pairwise difference of ASP4345 50 mg vs placebo) * sqrt(1/n[PLACEBO] + 1/n[ASP4345]). The Cohen's d Effect Size value for ASP4345 50 mg vs placebo is 0.035
Statistical Analysis 2: Comparison: Placebo vs ASP4345 150 mg; MMRM analysis model is performed with change from baseline (LS Mean estimate for observed value from separate model using observed values) at week 12 as response; treatment, site (pooled where necessary), visit, treatment*visit, and visit*baseline as fixed effects, and baseline as a covariate; Test type: Superiority; 0.775; LS Mean Difference = -0.28, 90% CI 2-sided [-1.93 to 1.36], Standard Error of Mean 0.99; Cohen's d Effect Size was defined as: (t-value for the least squares mean pairwise difference of ASP4345 150 mg vs placebo) * sqrt(1/n[PLACEBO] + 1/n[ASP4345]). The Cohen's d Effect Size value for ASP4345 150 mg vs placebo is - 0.053

2. Primary Outcome: Number of Participants With Adverse Event (AE)
Description: Treatment emergent adverse event (TEAE) is defined as an AE observed after starting administration of the study drug and 28 days after the last dose of study drug. A study drug-related TEAE is defined as any TEAE with at least possible relationship to study treatment as assessed by the investigator or with missing assessment of the causal relationship. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Safety was assessed by AEs, which included abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, metabolic parameters etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant.
Time Frame: Baseline up to end of study (EoS) (week 14)
Population: The safety analysis set (SAF) consisted of all participants who took at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | ASP4345 50 mg | ASP4345 150 mg
Number analyzed (Participants) | 100 | 65 | 68
participants
  TEAE | 45 | 28 | 28
  Drug-Related TEAEs | 11 | 13 | 11
  Serious TEAEs | 1 | 3 | 1
  Drug-Related Serious TEAE | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Differences in Columbia-Suicide Severity Rating Scale (C-SSRS) Values
Description: The C-SSRS is a questionnaire used for suicide risk assessment. Affirmative or negative responses are provided to items 1 to 5 for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods [not plan] without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and items 6 to 10 for suicide behavior (6. Preparatory acts or behavior, 7. Aborted attempt, 8. Interrupted attempt, 9. Actual attempt, 10. Completed suicide).
Time Frame: Baseline up to EoS (week 14)
Population: SAF population
Measure: Number; unit: participants
Arm/Group | Placebo | ASP4345 50 mg | ASP4345 150 mg
Number analyzed (Participants) | 100 | 65 | 68
participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Differences in Abnormal Involuntary Movement Scale (AIMS) Values
Description: AIMS is a 14-item scale. Items 1 to 8 are rated on a 5-point scale ranging from 0 (no dyskinetic movements) to 4 (severe dyskinetic movements). Item 9 assesses the participant's incapacitation due to abnormal movements, and item 10 assesses the participant's awareness of the abnormal movements and associated distress. Items 9 and 10 are rated on 5-point scales ranging from 0 (none or no awareness) to 4 (severe or aware, severe distress). Items 11 to 14 are yes/no questions regarding the global judgement and dental status of the participant. The total score is the sum of the scores for the 14 items and the possible total score ranges from 0 to 44. A higher total score is indicative of more severe dyskinetic movements.
Time Frame: Baseline, week 6 and week 12
Population: SAF population with available data at each time point.
Measure: Number; unit: participants
Arm/Group | Placebo | ASP4345 50 mg | ASP4345 150 mg
Number analyzed (Participants) | 93 | 62 | 65
participants
  Baseline | 0 | 0 | 0
  Week 6: number analyzed (Participants) | 83 | 55 | 60
  Week 6 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 70 | 46 | 52
  Week 12 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Differences in Simpson Angus Scale (SAS) Values
Description: SAS scale consists of 10 items including 7 items that address bradykinesia-rigidity and additional single items for tremor, glabellar tap, and salivation. Each item represents a specific physical condition and is rated on a 5-point category rating scale ranging from 0 (complete absence of the condition) to 4 (the condition is present to an extreme degree).The total score is obtained by adding the scores for the 10 individual items making the maximum possible score is 40. Higher scores are indicative of more severe Parkinsonian-type symptoms.
Time Frame: Baseline, week 6 and week 12
Population: SAF population with available data at each time point.
Measure: Number; unit: participants
Arm/Group | Placebo | ASP4345 50 mg | ASP4345 150 mg
Number analyzed (Participants) | 93 | 62 | 65
participants
  Baseline | 0 | 0 | 0
  Week 6: number analyzed (Participants) | 83 | 55 | 60
  Week 6 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 70 | 46 | 52
  Week 12 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Differences in Barnes Akathisia Rating Scale (BARS) Values
Description: BARS is used to rate observable, restless movements of drug induced akathisia and subjective awareness of restlessness and any distress associated with the akathisia. BARS consists of the following 4 items: objective assessment of akathisia symptoms, subjective assessment of the participants's awareness of inner restlessness, distress restlessness, and global clinical assessment of akathisia. First three items are rated on a 4-point scale ranging from 0 (no abnormal movements or absence of inner restlessness or no distress) to 3 (severe akathisia or awareness of intense compulsion to move most of the time or severe distress). The last item, the global clinical assessment of akathisia, is rated on a 6-point scale, ranging from 0 (no evidence of akathisia) to 5 (severe akathisia). Total BARS score ranges from 0 to 14 with a higher score representing worse results.
Time Frame: Baseline, week 6 and week 12
Population: SAF population with available data at each time point.
Measure: Number; unit: participants
Arm/Group | Placebo | ASP4345 50 mg | ASP4345 150 mg
Number analyzed (Participants) | 93 | 62 | 66
participants
  Baseline | 0 | 0 | 0
  Week 6: number analyzed (Participants) | 83 | 55 | 60
  Week 6 | 0 | 0 | 0
  Week 12: number analyzed (Participants) | 70 | 46 | 52
  Week 12 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline to Week 12/EoT in University of California San Diego Performance-based Skills Assessment-2 Extended Range (UPSA-2-ER) Total Score
Description: The UPSA-2-ER assesses the functional abilities of the participant with schizophrenia in 6 domains: household management, communication, financial skills, transportation, comprehension/planning and medication management. The UPSA-2-ER total score has a range from 0 to 105. A higher score indicates less impairment.
Time Frame: Baseline and week 12/EoT
Population: FAS population with available data at baseline and at week 12/EoT.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ASP4345 50 mg | ASP4345 150 mg
Number analyzed (Participants) | 55 | 40 | 44
units on a scale | 3.11 (1.06) | 3.86 (1.23) | 2.56 (1.17)
Statistical Analysis 1: Comparison: Placebo vs ASP4345 50 mg; Analysis of covariance (ANCOVA) model is performed with change from baseline (LS Mean estimate for observed value from separate model using observed values) at the Week 12 timepoint as response, treatment and site (pooled where necessary) and baseline as a covariate; Test type: Superiority; p = 0.639, ANCOVA; LS Mean Difference = 0.75, 90% CI 2-sided [-1.90 to 3.41], Standard Error of Mean 1.60
Statistical Analysis 2: Comparison: Placebo vs ASP4345 150 mg; ANCOVA model is performed with change from baseline (LS Mean estimate for observed value from separate model using observed values) at the Week 12 timepoint as response, treatment and site (pooled where necessary) and baseline as a covariate; Test type: Superiority; p = 0.721, ANCOVA; LS Mean Difference = -0.55, 90% CI 2-sided [-3.11 to 2.01], Standard Error of Mean 1.54

8. Secondary Outcome: Concentration at Trough Level (Ctrough) for ASP4345
Description: Ctrough concentration for ASP4345 was reported.
Time Frame: Predose: day 7, day 14, day 21, day 42 and day 84/EoT
Population: The pharmacokinetic analysis set (PKAS) consisted of all participants who took at least 1 dose of study drug and who had at least 1 plasma concentration. PKAS population with available data at each time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | ASP4345 50 mg | ASP4345 150 mg
Number analyzed (Participants) | 54 | 60
nanogram per milliliter (ng/mL)
  Day 7 Pre-dose | 175.041 (159.345) | 483.84 (452.65)
  Day 14 Pre-dose: number analyzed (Participants) | 48 | 49
  Day 14 Pre-dose | 182.903 (165.499) | 428.88 (516.14)
  Day 21 Pre-dose: number analyzed (Participants) | 15 | 17
  Day 21 Pre-dose | 172.040 (128.812) | 384.48 (331.71)
  Day 42 Pre-dose: number analyzed (Participants) | 46 | 44
  Day 42 Pre-dose | 207.145 (167.127) | 471.78 (546.00)
  Day 84 Pre-dose: number analyzed (Participants) | 35 | 39
  Day 84 Pre-dose | 204.914 (154.615) | 433.56 (427.12)

ADVERSE EVENTS:
Time Frame: Baseline up to EoS (week 14)
Arm/Group | Placebo | ASP4345 50 mg | ASP4345 150 mg
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/65 | 0/68
Serious Adverse Events (participants affected / at risk) | 1/100 | 3/65 | 1/68
Other Adverse Events (participants affected / at risk) | 3/100 | 5/65 | 7/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=100) | ASP4345 50 mg (N=65) | ASP4345 150 mg (N=68)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=100) | ASP4345 50 mg (N=65) | ASP4345 150 mg (N=68)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 3 (3) | 4 (4) | 3 (3)

LIMITATIONS AND CAVEATS:
ASP4345 metabolites were optional and deemed not necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT03557931/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03557931/SAP_001.pdf